CLINICAL TRIAL: NCT01594957
Title: An Open-label, Single Dose, Parallel-group Study to Evaluate the Pharmacokinetics of LCQ908 in Patients With Mild, Moderate and Severe Hepatic Impairment Compared to Age, Gender and Weight-matched Healthy Volunteers.
Brief Title: Pharmacokinetics of LCQ908 in Patients With Hepatic Impairment
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: CLCQ908B2101
Record Dates: First submitted 2012-05-07; First posted 2012-05-09 (Estimated); Last update posted 2020-12-19 (Actual); Status verified 2013-05

CONDITIONS: Hepatic Impairment
Keywords: LCQ908,; Hepatic Impairment,; Pharmacokinetics
MeSH Terms: interventions — pradigastat

ARMS (3):
- LCQ908 (mild hepatic impairment plus healthy volunteers) (Experimental): Healthy subjects will be matched pair-wise by, sex, race, age (±10 years) and weight (±20%) to subjects with mild hepatic impairment and will receive a single dose of LCQ908.
  Interventions: Drug: LCQ908
- LCQ908 (moderate hepatic impairment plus healthy volunteers) (Experimental): Healthy subjects will be matched pair-wise by, sex, race, age (±10 years) and weight (±20%) to subjects with moderate hepatic impairment and will receive a single dose of LCQ908.
  Interventions: Drug: LCQ908
- LCQ908 (severe hepatic impairment plus healthy volunteers) (Experimental): Healthy subjects will be matched pair-wise by, sex, race, age (±10 years) and weight (±20%) to subjects with severe hepatic impairment and will receive a single dose of LCQ908.
  Interventions: Drug: LCQ908

INTERVENTIONS:
Drug: LCQ908 — Participants will receive a single oral dose of LCQ908

SUMMARY:
This study will compare the pharmacokinetics of LCQ908 in subjects with varying degrees of hepatic impairment to healthy subjects.

ELIGIBILITY:
Inclusion criteria:

Individuals with hepatic impairment only

• Hepatic impairment evidenced by a Child-Pugh score

* Mild hepatic impairment defined Child-Pugh Class A (5-6 points)
* Moderate hepatic impairment defined Child-Pugh Class B (7-9 points)
* Severe hepatic impairment defined Child-Pugh Class C (10-15 points).

Healthy subjects only

• Good health determined.

Exclusion criteria:

All Individuals

* A past medical history of clinically significant ECG abnormalities or a family history of a prolonged QT-interval syndrome.
* Female subjects must be of non child bearing potential or use an effective method of contraception.

Individuals with hepatic impairment

* History of drug or alcohol abuse within 3 months prior to dosing.
* History or presence of significant uncontrolled disease of any major organ class.
* Any surgical or medical condition other than hepatic impairment which might alter the drug metabolism.

Healthy subjects

* History or presence of significant uncontrolled disease of any major organ class.
* Any surgical or medical condition other than hepatic impairment which might alter the drug metabolism.
* History or presence of hepatitis B or C and/or positive Hepatitis B surface antigen (HBsAg) or Hepatitis C test result at screening.

Other protocol-defined inclusion/exclusion criteria may apply.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2012-04; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Area under the plasma concentration-time profile from time zero to the time of the last quantifiable concentration (AUClast) of LCQ908 for part I of the study | Day 1 (treatment day) within 60 minutes prior to dosing, then, 1,2,4,6,8,10,12 hours after the dosing and on Days 2, 3, 4, 5, 6,7, 10, 13, 17, 21 and 28 post dosing
  This outcome applies to Part I of study involving mild and moderate hepatic impairment as well as healthy volunteers. Blood will be collected on Day 1 (treatment day) within 60 minutes prior to dosing, then, 1,2,4,6,8,10,12 hours after the dosing followed by additional blood draws on Days 2, 3, 4, 5, 6,7, 10, 13, 17, 21 and 28 post dosing.
Area under the plasma concentration-time profile from time zero extrapolated to infinite time [AUC(0-inf)] of LCQ908 for part I of the study | Day 1 (treatment day) within 60 minutes prior to dosing, then, 1,2,4,6,8,10,12 hours after the dosing and on Days 2, 3, 4, 5, 6,7, 10, 13, 17, 21 and 28 post dosing
  This outcome applies to Part I of study involving mild and moderate hepatic impairment as well as healthy volunteers. Blood will be collected on Day 1 (treatment day) within 60 minutes prior to dosing, then, 1,2,4,6,8,10,12 hours after the dosing followed by additional blood draws on Days 2, 3, 4, 5, 6,7, 10, 13, 17, 21 and 28 post dosing.
Maximum plasma concentration of LCQ908 (Cmax) for Part I of the study | Day 1 (treatment day) within 60 minutes prior to dosing, then, 1,2,4,6,8,10,12 hours after the dosing and on Days 2, 3, 4, 5, 6,7, 10, 13, 17, 21 and 28 post dosing
  This outcome applies to Part I of study involving mild and moderate hepatic impairment as well as healthy volunteers. Blood will be collected on Day 1 (treatment day) within 60 minutes prior to dosing, then, 1,2,4,6,8,10,12 hours after the dosing followed by additional blood draws on Days 2, 3, 4, 5, 6,7, 10, 13, 17, 21 and 28 post dosing.
The apparent systemic clearance (CL/F) of LCQ908 following extra vascular administration for Part I of the study | Day 1 (treatment day) within 60 minutes prior to dosing, then, 1,2,4,6,8,10,12 hours after the dosing and on Days 2, 3, 4, 5, 6,7, 10, 13, 17, 21 and 28 post dosing
  This outcome applies to Part I of study involving mild and moderate hepatic impairment as well as healthy volunteers. Blood will be collected on Day 1 (treatment day) within 60 minutes prior to dosing, then, 1,2,4,6,8,10,12 hours after the dosing followed by additional blood draws on Days 2, 3, 4, 5, 6,7, 10, 13, 17, 21 and 28 post dosing.
Area under the plasma concentration-time profile from time zero to the time of the last quantifiable concentration (AUClast) of LCQ908 for Part II of the study | Day 1 (treatment day) within 60 minutes prior to dosing, then, 1,2,4,6,8,10,12 hours after the dosing and on Days 2, 3, 4, 5, 6,7, 10, 13, 17, 21 and 28 post dosing
  This outcome applies to Part I of study involving mild and moderate hepatic impairment as well as healthy volunteers. Blood will be collected on Day 1 (treatment day) within 60 minutes prior to dosing, then, 1,2,4,6,8,10,12 hours after the dosing followed by additional blood draws on Days 2, 3, 4, 5, 6,7, 10, 13, 17, 21 and 28 post dosing.
Area under the plasma concentration-time profile from time zero extrapolated to infinite time [AUC(0-inf)] of LCQ908 for Part II of the study | Day 1 (treatment day) within 60 minutes prior to dosing, then, 1,2,4,6,8,10,12 hours after the dosing and on Days 2, 3, 4, 5, 6,7, 10, 13, 17, 21 and 28 post dosing
  This outcome applies to Part I of study involving mild and moderate hepatic impairment as well as healthy volunteers. Blood will be collected on Day 1 (treatment day) within 60 minutes prior to dosing, then, 1,2,4,6,8,10,12 hours after the dosing followed by additional blood draws on Days 2, 3, 4, 5, 6,7, 10, 13, 17, 21 and 28 post dosing.
Maximum plasma concentration of LCQ908 (Cmax) for Part II of the study | Day 1 (treatment day) within 60 minutes prior to dosing, then, 1,2,4,6,8,10,12 hours after the dosing and on Days 2, 3, 4, 5, 6,7, 10, 13, 17, 21 and 28 post dosing
  This outcome applies to Part I of study involving mild and moderate hepatic impairment as well as healthy volunteers. Blood will be collected on Day 1 (treatment day) within 60 minutes prior to dosing, then, 1,2,4,6,8,10,12 hours after the dosing followed by additional blood draws on Days 2, 3, 4, 5, 6,7, 10, 13, 17, 21 and 28 post dosing.
The apparent systemic clearance (CL/F) of LCQ908 following extra vascular administration for Part II of the study | Day 1 (treatment day) within 60 minutes prior to dosing, then, 1,2,4,6,8,10,12 hours after the dosing and on Days 2, 3, 4, 5, 6,7, 10, 13, 17, 21 and 28 post dosing
  This outcome applies to Part I of study involving mild and moderate hepatic impairment as well as healthy volunteers. Blood will be collected on Day 1 (treatment day) within 60 minutes prior to dosing, then, 1,2,4,6,8,10,12 hours after the dosing followed by additional blood draws on Days 2, 3, 4, 5, 6,7, 10, 13, 17, 21 and 28 post dosing.

SECONDARY OUTCOMES:
Number of participants with adverse events, serious adverse events and death (for both Part I and Part II) | Day 28
  Adverse events are defined as any unfavorable and unintended diagnosis, symptom, sign (including an abnormal laboratory finding), syndrome or disease which either occurs during study, having been absent at baseline, or, if present at baseline, appears to worsen. Serious adverse events are any untoward medical occurrences that result in death, are life threatening, require (or prolong) hospitalization,cause persistent or significant disability/incapacity, result in congenital abnormalities or birth defects,or are other conditions which in judgment of investigators represent significant hazards.
Time to maximum plasma concentration of LCQ908 (Tmax) (for both Part I and Part II) | Day 1 (treatment day) within 60 minutes prior to dosing, then, 1,2,4,6,8,10,12 hours after the dosing and on Days 2, 3, 4, 5, 6,7, 10, 13, 17, 21 and 28 post dosing
  This outcome applies to Part I and II of the study involving mild and moderate hepatic impairment as well as healthy volunteers for Part I, severe hepatic impairment and healthy volunteers for Part II. Blood will be collected on Day 1 (treatment day) within 60 minutes prior to dosing, then, 1,2,4,6,8,10,12 hours after the dosing and on Days 2, 3, 4, 5, 6,7, 10, 13, 17, 21 and 28 post dosing
The time required for the concentration of the drug to reach half of its original value (T1/2) (for both Part I and Part II) | Day 1 (treatment day) within 60 minutes prior to dosing, then, 1,2,4,6,8,10,12 hours after the dosing and on Days 2, 3, 4, 5, 6,7, 10, 13, 17, 21 and 28 post dosing
  This outcome applies to Part I and II of the study involving mild and moderate hepatic impairment as well as healthy volunteers for Part I, severe hepatic impairment and healthy volunteers for Part II. Blood will be collected on Day 1 (treatment day) within 60 minutes prior to dosing, then, 1,2,4,6,8,10,12 hours after the dosing and on Days 2, 3, 4, 5, 6,7, 10, 13, 17, 21 and 28 post dosing
The apparent volume of distribution of LCQ908 during the terminal elimination phase following extra vascular administration (Vz/F) (for both Part I and Part II) | Day 1 (treatment day) within 60 minutes prior to dosing, then, 1,2,4,6,8,10,12 hours after the dosing and on Days 2, 3, 4, 5, 6,7, 10, 13, 17, 21 and 28 post dosing
  This outcome applies to Part I and II of the study involving mild and moderate hepatic impairment as well as healthy volunteers for Part I, severe hepatic impairment and healthy volunteers for Part II. Blood will be collected on Day 1 (treatment day) within 60 minutes prior to dosing, then, 1,2,4,6,8,10,12 hours after the dosing and on Days 2, 3, 4, 5, 6,7, 10, 13, 17, 21 and 28 post dosing
LCQ908 protein binding: unbound area under curve (AUCu) of LCQ908 (for both Part I and Part II) | 10 and 24 hours post dose
  This outcome applies to Part I and II of the study involving mild and moderate hepatic impairment as well as healthy volunteers for Part I, severe hepatic impairment and healthy volunteers for Part II. Blood will be collected 10 and 24 hours post dosing.
LCQ908 protein binding: unbound observed maximum plasma (Cmax) of LCQ908 (for both Part I and Part II) | 10 and 24 hours
  This outcome applies to Part I and II of the study involving mild and moderate hepatic impairment as well as healthy volunteers for Part I, severe hepatic impairment and healthy volunteers for Part II. Blood will be collected 10 and 24 hours post dosing.
LCQ908 protein binding: unbound apparent systemic clearance from plasma (CL/Fu) following extra vascular administration (for both Part I and Part II) | 10 and 24 hours
  This outcome applies to Part I and II of the study involving mild and moderate hepatic impairment as well as healthy volunteers for Part I, severe hepatic impairment and healthy volunteers for Part II. Blood will be collected 10 and 24 hours post dosing.

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (2):
- United States (2):
  - Novartis Investigative Site, Miami, Florida
  - Novartis Investigative Site, Orlando, Florida

REFERENCES:
- [Derived] Hirano M, Meyers D, Golla G, Pal P, Pinot P, Lin T, Majumdar T, Rebello S, Sunkara G, Chen J. Effect of Hepatic Impairment on the Pharmacokinetics of Pradigastat, a Diacylglycerol Acyltransferase 1 (DGAT1) Inhibitor. Clin Pharmacokinet. 2015 Jul;54(7):761-70. doi: 10.1007/s40262-015-0235-9. PMID 25633714
- See also: Results for CCLCQ908B2101 can be found on the Novartis Clinical Trial Results Website — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=11443